CLINICAL TRIAL: NCT03426202
Title: The Effect of Modafinil on Neural Processing During the Interference and Feedback Based Learning Task
Brief Title: The Effect of Modafinil on Affective and Cognitive Processing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-49
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: modafinil; emotion; cognitive processing
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modafinil group (Experimental): a single dose of p.o. modafinil (200mg)
  Interventions: Drug: Modafinil Oral Tablet
- placebo group (Experimental): a single dose of p.o. placebo (200mg)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Modafinil Oral Tablet — modafinil 200mg
  Arms: modafinil group
Drug: Placebo Oral Tablet — placebo 200mg
  Arms: placebo group

SUMMARY:
The study aims to examine whether a single dose of modafinil (200mg, p.o.) can affect feedback-based learning and interference processing in healthy male subjects.

DETAILED DESCRIPTION:
Based on previous animal and human research suggesting a catecholamine-mediated, potentially pro-cognitive, mechanism of action of modafinil, the present study seeks to explore effects of modafinil on feedback-based learning and interference processing in healthy subjects. To this end, the present randomized double-blind, between-subject, placebo-controlled pharmaco-fMRI experiment plans to determine the behavioral and neural effects of a single dose of p.o.modafinil (200mg) versus placebo on validated feedback-based learning and emotional/non-emotional cognitive conflict paradigms. To control for potential effects of pre-medication personality traits as well as effects of modafinil on subjective task performance, subjects will be administered pre-treatment assessing relevant personality traits and post-treatment assessments of meta-cognitive confidence estimation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Non-smokers
* Right-handedness

Exclusion Criteria:

* Medical or psychiatric illness
* Allergy against medications or general strong allergies
* Sleep disorders
* High blood pressure, general cardio-vascular alterations
* History of head injury
* Visual or motor impairments

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Neural processing during the interference processing | 4h after treatment
  fMRI BOLD indices of neural processing in interference related brain regions will be compared between the treatment and placebo group.
Neural processing during feedback based learning | 4h after treatment
  fMRI BOLD indices of neural processing learning related brain regions will be compared between the treatment and placebo group.

SECONDARY OUTCOMES:
Behavioral interference performance - Response Time | 4h after treatment
  Behavioral performance of interference performance for congruent and incongruent stimuli (picture vs word) will be compared between the treatment and placebo group.
Behavioral interference performance - Accuracy | 4h after treatment
  Behavioral performance of interference in terms of accuracy for congruent and incongruent trials (picture vs word) will be compared between the treatment and placebo group.
Behavioral learning performance - Reaction time | 4h after treatment
  Learning performance in terms of reaction times will be compared between the treatment and placebo group.
Behavioral learning performance - Accuracy | 4h after treatment
  Learning performance in terms of accuracy (learning curve, trials to reach plateau) will be compared between the treatment and placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No